CLINICAL TRIAL: NCT04771598
Title: EVALUATING THE EFFICIENCY OF BREATHING EXERCISES PERFORMED BY POST-COVID TELEMEDICINE: Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Fatih OKAN, Assist. Prof., Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 123458
Record Dates: First submitted 2021-02-21; First posted 2021-02-25 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention (Experimental): Respiratory exercises will be instructed to the individuals forming the intervention group and participants will be asked to do 3 times a day during one month and the exercises will be done by the researchers together with the individuals by establishing a connection with the phone application (zoom, watsapp) once a week from home. In terms of physical activity, the patient will be encouraged to participate in the program by suggesting exercises such as walking and cycling at least three times a week for 20 minutes per week
  Interventions: Other: Breathing exercise with the phone application
- Control (Other): Breathing exercises will be explained to the control group and visual material will be given. The participants will be asked to do 3 times a day during one month. In terms of physical activity, the patient will be encouraged to participate in the program by suggesting exercises such as walking and cycling at least three times a week for 20 minutes per week
  Interventions: Other: Breathing exercise

INTERVENTIONS:
Other: Breathing exercise with the phone application — 1. Respiratory Control:
  2. Pursed Lip Breathing
  3. Diaphragmatic Breathing Respiratory exercises will be instructed to the individuals forming the intervention group and participants will be asked to do 3 times a day during one month and the exercises will be done by the researchers together with the individuals by establishing a connection with the phone application (zoom, watsapp) once a week from home.
  Arms: İntervention
Other: Breathing exercise — 1. Respiratory Control:
  2. Pursed Lip Breathing
  3. Diaphragmatic Breathing Breathing exercises will be explained to the control group and visual material will be given. The participants will be asked to do 3 times a day during one month. In terms of physical activity, the patient will be encouraged to participate in the program by suggesting exercises such as walking and cycling at least three times a week for 20 minutes per week
  Arms: Control

SUMMARY:
As an important non-drug intervention in the treatment of respiratory tract diseases, respiratory rehabilitation training is increasingly accepted in clinical practice. The purpose of pulmonary rehabilitation is not only to improve the physical and mental conditions of the patient, but also to help the patient return to the family and society more quickly.

In light of the widely documented lung injuries associated with COVID-19, concerns are raised regarding the assessment of lung injury in discharged patients. As an important non-drug intervention in the treatment of respiratory diseases, respiratory rehabilitation training is increasingly being accepted in clinical practice The purpose of pulmonary rehabilitation is not only to improve the physical and mental conditions of the patient, but also to help the patient return to the family and society more quickly.

The aim of the study; It is aimed to evaluate the efficiency of breathing exercise in individuals with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older and who received / will receive treatment with the diagnosis of COVID 19 and completed 2 months after the diagnosis of COVID 19
* Patients who applied to the Pulmonary Diseases outpatient clinic with complaints of dyspnea
* FEV1 / FVC <80%, FVC <80%, FEV1 <80%, FEF25-75> 50% and / or Patients with respiratory distress in daily living activities

Exclusion Criteria:

* FEV 1 <50%, FEF 25-75 <50% detected oxygen saturation <85% at rest,
* moderately severe heart failure,
* has a disease that restricts its mobilization,
* psychiatric illness,
* advanced stage liver, advanced stage renal failure,
* Myocardial infarction within 4 months
* having a history of unstable angina
* active infectious disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
6 minute walking test | 1 month
  6 minute walking test
FEV-1 | 1 month
  FEV-1
FVC | 1 month
  FVC
FEV1/FVC | 1 month
  FEV1/FVC
MVV | 1 month
  MVV- Maximal Voluntary Ventilation

SECONDARY OUTCOMES:
St. George's Respiratory Questionnaire | 1 month
  St. George's Respiratory Questionnaire-Scores range from 0 to 100, with higher scores indicating more limitations.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat State Hospital, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No